CLINICAL TRIAL: NCT05887167
Title: IIT2022-04-Sasine-CAR-T: A Phase 1 Single-arm, Open-label Study to Evaluate the Feasibility and Safety of Collecting and Combining Autologous Hematopoietic Stem Cells With Chimeric Antigen Receptor (CAR) T-Cell Therapy in Subjects With Relapsed/Refractory Hematological Malignancies
Brief Title: Feasibility and Safety of Collecting and Combining Autologous Hematopoietic Stem Cells With Chimeric Antigen Receptor (CAR) T-Cell Therapy in Subjects With Relapsed/Refractory Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joshua Sasine, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joshua Sasine, MD, PhD, Assistant Professor of Medicine, Co-Director, CAR T Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022-04-Sasine-CAR-T
Record Dates: First submitted 2023-05-17; First posted 2023-06-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy; Large B-cell Lymphoma; Acute Lymphoblastic Leukemia; Mantle Cell Lymphoma; Multiple Myeloma; Diffuse Large B Cell Lymphoma
Keywords: CAR T-cell therapy; autologous hematopoietic stem cells; CAR T; CAR T therapy
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR T Therapy with Autologous Hematopoietic Stem Cells (aHSCs) (Experimental)
  Interventions: Biological: autologous hematopoietic stem cells added to planned CAR T

INTERVENTIONS:
Biological: autologous hematopoietic stem cells added to planned CAR T — Autologous hematopoietic stem cells (aHSCs) infused on Day 10 after CAR T (any FDA-approved CAR T product) infusion on Day 0.

SUMMARY:
The study is designed to examine the feasibility and safety of collecting autologous hematopoietic stem cells (HSCs) to be combined with CAR T-cell therapy for patients with relapsed/refractory (r/r) hematological disease. The study will evaluate feasibility of collecting the target dose of HSCs from at least 50% of enrolled patients. The study will assess safety based on incidence and severity of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) in the first 60 days post CAR T dosing, and also through the collection of adverse events (AEs) and serious adverse events (SAEs) as well as the durability of response after treatment with HSCs with CAR T. The study follows an open-label, single-center and single non-randomized cohort design. 20 subjects with r/r hematological malignancies will be enrolled and treated to evaluate the feasibility and preliminary safety of collecting autologous HSCs and combining them with CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years.
* Histologically proven hematological malignancy according to the World Health Organization 2016 classification criteria for which a commercially available, FDA-approved CAR T product exists.
* Relapsed or refractory disease, defined by the following:

  * Disease progression after last regimen, or
  * Refractory disease: failure to achieve a partial response (PR) or complete remission (CR) to the last regimen
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy for the malignancy at the time the subject is planned for leukapheresis.
* Toxicities due to prior therapy must be stable or recovered to ≤ Grade 1 with the exception of alopecia.
* Subjects with an active uncontrolled infection should not start CAR T treatment until the infection has resolved.
* Eastern cooperative oncology group (ECOG) performance status 0 - 2.
* Adequate hematologic, hepatic, and cardiac function
* Serum pregnancy test for women of childbearing potential (WOCBP) at Screening.
* Willing to comply to research specimen collection as specified in the protocol.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Autologous hematopoietic cell transplant intent or execution within 8 weeks of planned CAR T infusion.
* History of allogeneic cell transplantation within 8 weeks of planned CAR T infusion.
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management at time of screening.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment.
* History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, or any autoimmune disease with CNS involvement.
* Doses of corticosteroids of greater than or equal to 5 mg/day of prednisone or equivalent doses of other corticosteroids and other immunosuppressive drugs are not allowed prior to enrollment. A washout period of 10 days prior to leukapheresis and 10 days prior to anti-CD19 CAR T cell administration is required.
* Any medical condition likely to interfere with assessment of feasibility or safety of study treatment.
* Live vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Current pregnancy or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Subjects of both sexes who are not willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females who have undergone surgical sterilization or who have been postmenopausal for at least 1 year are not considered to be of childbearing potential.
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
* Patients with obvious myeloid clonal hematopoiesis on the screening bone marrow biopsy will be excluded based on the risk of developing myeloid neoplasms with aHSC infusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility of collecting the target HSC cell dose for at least 50% of enrolled patients. | From Day 0 (CAR T infusion) to Day 10 (aHSC infusion).
  Target dose collection of autologous HSCs (2 to 5 x 106 CD34+ cells/kg) defined as collection from at least 50% of patients enrolled in this study by Day 10.
To assess safety of aHSC to planned CAR T therapy in the first 60 days through the incidence, severity, and duration of CRS based on the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading system. | From Day 0 to Day 60.
  Safety will be assessed by incidence, severity, and duration of CRS per ASTCT consensus grading system. ASTCT CRS Consensus grading (Grade scale is 1-4) is based on 3 CRS parameters: fever, hypotension, and hypoxia. Higher grade indicates worse outcome.
To assess safety of aHSC to planned CAR T therapy in the first 60 days through the incidence, severity, and duration of ICANS based on the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading system. | From Day 0 to Day 60.
  Safety will be assessed by incidence, severity, and duration ICANS per ASTCT consensus grading system. ASTCT ICANS Consensus grading (Grade scale is 1-4) is based on 5 neurotoxicity domains: Immune Effector Cell-Associated Encephalopathy (ICE) score, level of consciousness, seizure, motor findings, raised intracranial pressure (ICP)/cerebral edema. Higher grade indicates worse outcome.

SECONDARY OUTCOMES:
Response rate of CAR T at 6 weeks. | From Day 0 to Day 60.
  Response rate of CAR T will be defined as the proportion of subjects who experience partial response (PR) or complete response (CR) assessed at 6 weeks or day 60. Response criteria used will be according to type of disease: Response by International Myeloma Working Group (IMWG) Criteria (for multiple myeloma); Response by Center for International Blood and Marrow Transplant Research (CIMBTR) Criteria (for acute lymphoblastic leukemia); Response by Lugano Criterial (for lymphoma).
Assess rate of recovery of absolute neutrophil count (ANC) by Day 28. | From Day 0 to Day 28.
  Recovery assessed by the proportion of patients with ANC recover to ≥ 500/µL.
Assess red blood cell (RBC) count and transfusion independence by Day 28. | From Day 0 to Day 28.
  The proportion of patients with RBC transfusion independence by Day 28.
Assess platelet count and transfusion independence rate by Day 28. | From Day 0 to Day 28.
  The proportion of patients with platelet transfusion independence by Day 28.
Assess safety and tolerability of combining aHSCs with an FDA-approved CAR T regimen within first 52 weeks of aHSC infusion. | From Day 0 to Week 52.
  Safety and tolerability will be assessed by the number of adverse events (AEs) and serious adverse events (SAEs) related to study treatment according to CTCAE v.5, up to Week 52.
Median progression-free survival (PFS) for the duration of the study | From Day 0 until disease progression or withdrawal. Assessed up to 3 years.
  PFS will be assessed from time of CAR T infusion until confirmation of disease progression or withdrawal of consent, whichever comes first.
Median overall survival (OS) for the duration of the study | From Day 0 until death due to any cause or withdrawal of consent. Assessed up to 3 years.
  OS will be assessed from date of CAR T infusion until date of death due to any cause or withdrawal of consent, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Sasine, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No